CLINICAL TRIAL: NCT03927079
Title: Predictive Factors of Good Pulmonary Penetration of Antibiotics : AntiBiotics Dosage in Broncho-Alveolar Lavage
Acronym: ABBA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2018_843_0032
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Antibiotics; Pneumonia
Keywords: Antibiotics; Pneumonia; broncho-alveolar lavage
MeSH Terms: conditions — Pneumonia | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: measure of intra-alveolar antibiotic concentration in µg/ml — included patients will have a broncho-alveolar lavage (BAL) to measure intra-alveolar antibiotic concentration, and a blood test to measure plasmatic concentration
Procedure: broncho-alveolar lavage (BAL) — included patients will have a broncho-alveolar lavage (BAL) to measure intra-alveolar antibiotic concentration, and a blood test to measure plasmatic concentration
Biological: blood test to measure plasmatic antibiotic concentration in µg/ml — included patients will have a broncho-alveolar lavage (BAL) to measure intra-alveolar antibiotic concentration, and a blood test to measure plasmatic

SUMMARY:
Respiratory infections are common and sometimes very severe. An insufficient dosage of the antibiotic could lead to a treatment failure A correct plasmatic antibiotic concentration is not a guarantee of a clinical success as it could not be a reflect of pulmonary concentration. The aim of this study is to determinate the predictive factors of pulmonary penetration of antibiotics in patients with a beta lactamines failure and who undergoes a flexible bronchoscopy.

DETAILED DESCRIPTION:
To check if pulmonary concentrations of antibiotic are enough we will measure antibiotic concentration in the broncho-alveolar lavage (BAL). This technique which is clinically relevant and reliable could determinate the pulmonary diffusion level for antibiotics by calculating the ratio between plasmatic and intra-alveolar antibiotic concentration. This ratio will be correlated with potential limitation factors of pulmonary diffusion as respiratory diseases (COPD, cystic fibrosis, fibrosis…), sepsis, hypoalbuminemia. We have chosen to study the beta lactamin antibiotics because they are the most frequently used in pneumonia. Moreover, the beta lactamins pulmonary diffusion is likely to be the lowest. Finally, for patients with a known pathogen, we will divide this pulmonary concentration with minimal inhibitory concentration (MIC). Indeed, in severe pneumonia, to be sure of bactericidal activity, a pulmonary concentration of beta lactamines should be always higher than 4 to 5 times MIC.

ELIGIBILITY:
Inclusion Criteria:

* patients who undergo a flexible bronchoscopic lavage and with a beta lactamines treatment as cephalosporin of 3rd generation (CEFTRIAXONE / CEFOTAXIME, CEFTAZIDIME), of 4th generation (CEFEPIM), or AMOXICILLIN-CLAVULANIC ACID, or PIPERACILLIN-TAZOBACTAM
* patient major
* informed and signed consent form

Exclusion Criteria:

* patient under chronic dialysis
* patient placed under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
pulmonary diffusion level for beta lactamins | on the day of the bronco-alveolar lavage
  pulmonary diffusion level for beta lactamins is determined by ratio between bronchoalveolar concentration and plasmatic concentration of tested antibiotics

SECONDARY OUTCOMES:
measure of apyrexia duration in days | from day of inclusion to 15 days after inclusion
  measure of apyrexia duration in days
duration in days for regression of the biological inflammatory syndrome | from day of inclusion to 15 days after inclusion
  duration in days for regression of the biological inflammatory syndrome (CRP concentration in mg/l divided by 2)
measure of length of hospitalisation | from day of inclusion to 15 days after inclusion
  measure of length of hospitalisation in days
Number of deaths at 28-day | 28 days after inclusion
  28-day mortality will be measured
virus presence in BAL | day of bronchoalveolar lavage (BAL)
  virus presence will be detected in bronchoalveolar lavage (BAL)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Andrejak, Pr, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No